CLINICAL TRIAL: NCT00199420
Title: A 12-week, Double Blind, Placebo-controlled, Randomized, Parallel Group, Multicenter, Fixed Dose Study to Evaluate the Efficacy and Safety of 10, 20 and 40 mg/d Oral Dose of KW-6002 (Istradefylline) as Treatment for Parkinson's Disease in Patients With Motor Response Complications on Levodopa/Carbidopa Therapy.
Brief Title: A Study of Istradefylline (KW-6002) in Treating Patients With Parkinson's Disease on Levodopa
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kyowa Kirin, Inc. (Industry)
Organization: Kyowa Kirin Co., Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 6002-US-018; NCT00203983 (obsolete NCT alias)
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Parkinson's Disease
Keywords: levodopa; end of dose wearing off; OFF time
MeSH Terms: conditions — Parkinson Disease | interventions — istradefylline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Istradefylline (KW-6002)

SUMMARY:
To establish the efficacy of 10, 20 and 40 mg/d dose of istradefylline for reducing the percentage of OFF time in patients with advanced Parkinson's disease (PD) treated with levodopa.

DETAILED DESCRIPTION:
To establish the efficacy of 10, 20 and 40 mg/d dose of istradefylline for reducing the percentage of OFF time in patients with advanced Parkinson's disease (PD) treated with levodopa. Patients who meet entry criteria will be randomized in a 1 to 1 ratio to either istradefylline 10, 20 or 40 mg or matching placebo. Patients will be treated for 12 weeks and will have interim visits and end of treatment visit to assess efficacy and safety.

ELIGIBILITY:
Inclusion Criteria:

1. UK Parkinson's Disease Society (UKPDS) brain bank criteria (Step 1 and 2) for PD.
2. PD stages 2-4 in the OFF state for Modified Hoehn and Yahr Scale.
3. On levodopa/carbidopa for at least one year, stable dose in past 4 weeks.
4. Currently take at least three doses of levodopa/carbidopa per day.
5. Predictable end of dose wearing off.
6. Able to satisfactorily complete Hauser version of a Parkinson's diary.
7. Have an average of 180 minutes of OFF time on two 24 hour diaries.
8. Be at least 30 years of age.

Exclusion Criteria:

1. Neurosurgical treatment for PD.
2. History of psychosis.
3. Diagnosis of atypical parkinsonism, secondary parkinsonism variant or Parkinson's plus syndromes.
4. Diagnosis of cancer within 5 years.
5. Mini-mental status examination score of 25 or less.
6. History of seizures or neurologic malignant_syndrome.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 580
Dates: Start 2004-07; Primary Completion 2005-11 (Actual); Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
To establish the efficacy of 10, 20 and 40 mg/d istradefylline for reducing the percentage of OFF time in patients with advanced Parkinson's disease (PD) treated with levodopa/carbidopa.

SECONDARY OUTCOMES:
To evaluate the dose-response of 10, 20 and 40 mg/d istradefylline using the primary efficacy outcome variable.
To evaluate the efficacy of 10, 20 and 40 mg/d istradefylline for reducing the total hours of OFF time.
To evaluate the change in total hours of ON time (without dyskinesia, with dyskinesia, with non-troublesome dyskinesia, and with troublesome dyskinesia).
To evaluate the change in Unified Parkinson's Disease Rating Scale (UPDRS) Motor Examination score (part III) and/or in Activities of Daily Living (ADL) score (part II).
To evaluate the change in Parkinson's Disease Questionnaire (PDQ-39) and Medical Outcomes Study 36-item Short Form (SF-36).
To evaluate the Patient Global Impression - Improvement scale (PGI-I).
To evaluate change in the Clinical Global Impression - Severity of Illness scale (CGI-S).
To evaluate the safety of 10, 20, and 40 mg/d istradefylline by changes in safety parameters as noted in Section 7.2.4.

CONTACTS AND LOCATIONS:
Overall Officials: Neil Sussman, MD, Study Director — Kyowa Kirin, Inc.
Locations (2):
- United States (2):
  - Kyowa Pharmaceutical Inc., Princeton, New Jersey
  - Kyowa Pharmaceutical, Princeton, New Jersey